CLINICAL TRIAL: NCT04789902
Title: A Stepped Wedge Cluster Randomized Trial Designed to Evaluate the Effects of SurgeCon: A Quality Improvement Surge Management Platform
Brief Title: SurgeCon: An Emergency Department Surge Management Platform
Acronym: SurgeCon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Government of Newfoundland and Labrador (Other Government); Eastern Health (Other); Trinity Conception Placentia Health Foundation (Unknown)
Responsible Party: Principal Investigator, Shabnam Asghari, Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20201482; SR4-165123 (Other Grant/Funding Number: CIHR and other local provincial sponsors)
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Length of Stay; Emergency Departments
Keywords: SurgeCon; Emergency Department; Stepped-Wedge Design; Randomized Trials; Wait Time
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomized trial (SW-CRT) design, where the sequential crossover will occur in one direction. SW-CRT is a flexible CRT design progressively being used in trial arms with varying delays in switching from the control condition to the active intervention condition state. This study will include the implementation of the intervention in four different rural and urban hospitals. Therefore, one hospital will be randomly allocated using a stratified sampling technique to each of four sequences, which will determine the order in which the intervention is implemented across participating hospitals or clusters. This allocation of one cluster to each sequence maximizes the statistical power
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hospital site 1 (Experimental): This site will provide usual ED care during the control period which will last for the first six months of the study. After six months this site will begin transitioning to the SurgeCon management platform which they will use until the end of the study.
  Interventions: Other: SurgeCon
- Hospital site 2 (Experimental): This site will provide usual ED care during the control period which will last for the first 12 months of the study. After 12 months this site will begin transitioning to the SurgeCon management platform which they will use until the end of the study.
  Interventions: Other: SurgeCon
- Hospital site 3 (Experimental): This site will provide usual ED care during the control period which will last for the first 18 months of the study. After 18 months this site will begin transitioning to the SurgeCon management platform which they will use until the end of the study.
  Interventions: Other: SurgeCon
- Hospital site 4 (Experimental): This site will provide usual ED care during the control period which will last for the first 24 months of the study. After 24 months this site will begin transitioning to the SurgeCon management platform which they will use until the end of the study.
  Interventions: Other: SurgeCon

INTERVENTIONS:
Other: SurgeCon — The SurgeCon intervention is a pragmatic ED management platform that includes three distinct intervention components which include 1) Restructuring ED Organization & Workflow, 2) Establishing a Patient-Centric ED Environment, and 3) E-Health Action-Based ED Management that together act to improve ED efficiency and patient satisfaction and value of care.

SUMMARY:
Wait times and overcrowding are challenging emergency departments (EDs) around the world. Several countries with advanced healthcare systems cannot keep pace with patient demand, and Canada ranks among the longest wait times compared to peer-industrialized countries. In fact, the Canadian Institute for Health Information (CIHI) identified an 11% increase in ED wait times from 2015-2016 to 2016-2017. This translates to long wait times that deter patients from pursuing necessary care and increases their likelihood of leaving without being seen by an ED physician. In Newfoundland and Labrador (NL), this issue has precipitated strikingly serious situations regarding long wait times that have made the province a case-in-point for ED issues. To counter this, the investigators propose an innovative quality-improvement intervention called SurgeCon that includes a protocol-driven software platform and several other initiatives to reduce wait times and improve the sustainability of health systems without significant workforce changes. The investigators piloted SurgeCon at the ED in Carbonear, Newfoundland and Labrador (NL) and found there was a 32% reduction in ED wait time.

DETAILED DESCRIPTION:
Emergency Department (ED) wait times and overcrowding is a national problem of considerable magnitude with few favorable solutions. Canadian EDs are failing to meet national targets and have some of the longest wait times compared to peer industrialized countries. For patients, long wait times mean pain or discomfort for hours before being seen. To address these challenges, the investigators propose "SurgeCon", a quality improvement platform to reduce ED wait times and improve patient satisfaction. This study will investigate the effects of SurgeCon on health system key performance outcomes and patient-reported experience and satisfaction. The study uses a comparative effectiveness-implementation hybrid design. This type of hybrid design has been recommended to help achieve rapid translational gains that can hasten the movement of interventions from research to practice to public health impact. In our hybrid design, the investigators will use a pragmatic stepped wedge cluster randomized trial (SW-CRT) design that enrols four 24/7 on-site ED physician support (category A) hospitals into a 31-month trial. At the beginning of the trial, participating sites will operate under a 'usual care' model as a control condition. Each site will transition from providing 'usual care' to the new 'care model' at predetermined periods during the study. At the end of the trial, each of the sites will have eventually transitioned to the SurgeCon enabled care model. Each cluster in this trial will be randomly assigned to an arm of the trial as is the case with most stepped wedge trials.

The platform includes an eHealth component, a training program for ED staff, and a series of quality improvement initiatives. SurgeCon optimizes patient flow and creates a more patient-centric environment; it monitors ED capacity in real-time and helps address overcrowding by prescribing a series of actions customized to maximize patient flow in response to the level of demand in the ED. SurgeCon was recently piloted in a rural hospital and was associated with dramatic improvements in ED efficiency. Our time series analysis showed a significant decrease in the number of patients who left the ED without being seen by a physician (LWBS) (12.1% to 4.6%, p<0.004), time to physician initial assessment (PIA) (104.3 minutes to 42.2 minutes, p<0.001), and length of stay in the ED (LOS) (199.4 minutes to 134.4 minutes p<0.002).

The investigators plan to implement and evaluate SurgeCon in other hospitals in Newfoundland and Labrador (NL) to determine whether these results can be reproduced in urban and other rural EDs. SurgeCon will be considered a completely successful intervention if it requires minimal resources from the ED/health system for its continued operation, improves patient satisfaction and outcomes, and creates better value ED services by reducing the cost of providing the services. The payer organization that will be a rewarding success is the Eastern Health regional health authority (EH) in NL. As the largest health authority in NL, EH is a key organization for the delivery of care and setting provincial standards. It is responsible for managing both rural and urban hospitals and reflects the diversity of institutions across the rest of Canada.

SurgeCon's evaluation and implementation strategy will include a four-stage iterative process: 1. Exploration (month 1-10); 2. Adoption (months 11-12, 17-18, 23-24 and 29-30); 3. Active Implementation (months 13-36); 4. Sustainment (months 19-48). To measure success, the investigators will use an innovative comparative effectiveness implementation hybrid design. The investigators will test the effects of SurgeCon on ED key performance indicators (LOS, PIA, and LWBS) and patient-reported experiences (PREMs), while also capturing data related to its implementation across participating EDs. Our innovative clinical trial (iCT) design will test the effectiveness of SurgeCon using a pragmatic stepped wedge cluster randomized controlled trial accompanied by a cost-effectiveness analysis. Our stepped-wedge iCT design will assign each hospital to a step through a random ordering process. In addition to ED key performance indicators (KPI) and PREMs, the investigators will also measure implementation outcomes related to SurgeCon's scalability, adaptability, sustainability and overall costs. Implementation outcomes will be evaluated by patients, providers/staff and health system managers using a mixed methods process. The hybrid evaluation/implementation design represents an integrated knowledge translation approach that will ensure research findings are eventually integrated into policy and practice. Moreover, a multidisciplinary research team including patient partners, decision-makers, frontline clinicians, and researchers will lead this research.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who visit any of the four selected emergency departments during the study period will be included.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436052 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 31 Months
  Key Performance Indicator (KPI) data at the time of the emergency department visit. Total length of stay in the emergency department. Patients are either admitted/transferred to an inpatient unit in the hospital or discharged from the emergency department.
Time to physician's initial assessment | 31 Months
  Key Performance Indicator (KPI) data at the time of the ED visit. Also referred to as 'door to doctor' time. It is the amount of time it takes from patient arrival to being seen by a physician or their delegate.
Number of patients left without being seen | 31 Months
  Key Performance Indicator (KPI) data at the time of the ED visit. Patients who are registered and/or triaged but leave before being seen by a physician or their delegate.

SECONDARY OUTCOMES:
Patient satisfaction and patient reported experiences with ED wait time | 31 Months
  Patient-reported experiences and patient satisfaction will be collected via telephone interviews with patients who will be contacted 3 to 5 days after ED/hospital discharge. The telephone interviews will be conducted by a research assistant who is also an Eastern Health employee.
Economic impact of intervention on emergency department services | 31 Months
  Cost of providing emergency department services (this includes but not limited to the cost of pharmacy, lab tests, diagnostic imaging, and therapeutic interventions).

CONTACTS AND LOCATIONS:
Overall Officials: Shabnam Shabnam, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (4):
- Canada (4):
  - Burin Peninsula Healthcare Centre, Burin, Newfoundland and Labrador
  - Dr. G.B. Cross Memorial Hospital, Clarenville, Newfoundland and Labrador
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available only for the people involved in data analysis. Reports generated by the analysis will be will only include aggregate level information and will be made available to other members of the research team and will be used for publications.

REFERENCES:
- [Background] Torjesen I. Latest waiting time figures for emergency departments in England are worse on record. BMJ. 2018 Apr 12;361:k1658. doi: 10.1136/bmj.k1658. No abstract available. PMID 29650511
- [Background] Vezyridis P, Timmons S. National targets, process transformation and local consequences in an NHS emergency department (ED): a qualitative study. BMC Emerg Med. 2014 Jun 13;14:12. doi: 10.1186/1471-227X-14-12. PMID 24927819
- [Background] Chang AM, Lin A, Fu R, McConnell KJ, Sun B. Associations of Emergency Department Length of Stay With Publicly Reported Quality-of-care Measures. Acad Emerg Med. 2017 Feb;24(2):246-250. doi: 10.1111/acem.13102. PMID 27640877
- [Background] Carter AJ, Chochinov AH. A systematic review of the impact of nurse practitioners on cost, quality of care, satisfaction and wait times in the emergency department. CJEM. 2007 Jul;9(4):286-95. doi: 10.1017/s1481803500015189. PMID 17626694
- [Background] Maggio PM, Brundage SI, Hernandez-Boussard T, Spain DA. Commitment to COT verification improves patient outcomes and financial performance. J Trauma. 2009 Jul;67(1):190-4; discussion 194-5. doi: 10.1097/TA.0b013e3181a51b2f. PMID 19590334
- [Background] Jarvis PR. Improving emergency department patient flow. Clin Exp Emerg Med. 2016 Jun 30;3(2):63-68. doi: 10.15441/ceem.16.127. eCollection 2016 Jun. PMID 27752619
- [Background] Schroeppel TJ, Sharpe JP, Magnotti LJ, Weinberg JA, Croce MA, Fabian TC. How to increase the burden on trauma centers: implement the 80-hour work week. Am Surg. 2014 Jul;80(7):659-63. PMID 24987896
- [Background] Schroeppel TJ, Sharpe JP, Magnotti LJ, Weinberg JA, Croce MA, Fabian TC. How to Further Decrease the Efficiency of Care at a Level I Trauma Center: Implement the Amended Resident Work Hours. Am Surg. 2015 Jul;81(7):698-703. PMID 26140890
- [Background] Christmas E, Johnson I, Locker T. The impact of 24 h consultant shop floor presence on emergency department performance: a natural experiment. Emerg Med J. 2013 May;30(5):360-2. doi: 10.1136/emermed-2012-201369. Epub 2012 Jun 1. PMID 22660466
- [Background] Han JH, Zhou C, France DJ, Zhong S, Jones I, Storrow AB, Aronsky D. The effect of emergency department expansion on emergency department overcrowding. Acad Emerg Med. 2007 Apr;14(4):338-43. doi: 10.1197/j.aem.2006.12.005. PMID 17400996
- [Background] Mumma BE, McCue JY, Li CS, Holmes JF. Effects of emergency department expansion on emergency department patient flow. Acad Emerg Med. 2014 May;21(5):504-9. doi: 10.1111/acem.12366. PMID 24842500
- [Background] van Veelen MJ, van den Brand CL, Reijnen R, van der Linden MC. Effects of a general practitioner cooperative co-located with an emergency department on patient throughput. World J Emerg Med. 2016;7(4):270-273. doi: 10.5847/wjem.j.1920-8642.2016.04.005. PMID 27942343
- [Background] Morin C, Choukroun J, Callahan JC. Safety and efficiency of a redirection procedure toward an out of hours general practice before admission to an emergency department, an observational study. BMC Emerg Med. 2018 Aug 22;18(1):26. doi: 10.1186/s12873-018-0173-6. PMID 30134934
- [Background] Barker D, McElduff P, D'Este C, Campbell MJ. Stepped wedge cluster randomised trials: a review of the statistical methodology used and available. BMC Med Res Methodol. 2016 Jun 6;16:69. doi: 10.1186/s12874-016-0176-5. PMID 27267471
- [Background] Beard E, Lewis JJ, Copas A, Davey C, Osrin D, Baio G, Thompson JA, Fielding KL, Omar RZ, Ononge S, Hargreaves J, Prost A. Stepped wedge randomised controlled trials: systematic review of studies published between 2010 and 2014. Trials. 2015 Aug 17;16:353. doi: 10.1186/s13063-015-0839-2. PMID 26278881
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Jiang, Jiming. "Consistent Estimators in Generalized Linear Mixed Models." Journal of the American Statistical Association, vol. 93, no. 442, 1998, pp. 720-729. JSTOR, www.jstor.org/stable/2670122. Accessed 2 Mar. 2021.
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Martin J, Taljaard M, Girling A, Hemming K. Systematic review finds major deficiencies in sample size methodology and reporting for stepped-wedge cluster randomised trials. BMJ Open. 2016 Feb 4;6(2):e010166. doi: 10.1136/bmjopen-2015-010166. PMID 26846897
- [Background] Kumar A, Chakraborty BS. Interim analysis: A rational approach of decision making in clinical trial. J Adv Pharm Technol Res. 2016 Oct-Dec;7(4):118-122. doi: 10.4103/2231-4040.191414. PMID 27833889
- [Background] Shippee ND, Domecq Garces JP, Prutsky Lopez GJ, Wang Z, Elraiyah TA, Nabhan M, Brito JP, Boehmer K, Hasan R, Firwana B, Erwin PJ, Montori VM, Murad MH. Patient and service user engagement in research: a systematic review and synthesized framework. Health Expect. 2015 Oct;18(5):1151-66. doi: 10.1111/hex.12090. Epub 2013 Jun 3. PMID 23731468
- [Background] Kamine TH, Rembisz A, Barron RJ, Baldwin C, Kromer M. Decrease in Trauma Admissions with COVID-19 Pandemic. West J Emerg Med. 2020 May 22;21(4):819-822. doi: 10.5811/westjem.2020.5.47780. PMID 32726250
- [Background] Vashi AA, Sheikhi FH, Nashton LA, Ellman J, Rajagopal P, Asch SM. Applying Lean Principles to Reduce Wait Times in a VA Emergency Department. Mil Med. 2019 Jan 1;184(1-2):e169-e178. doi: 10.1093/milmed/usy165. No abstract available. PMID 30007347
- [Background] Matthias H. The genealogy of lean production. Journal of Operations Management. 2007 2;25: doi.org/10.1016/j.jom.2006.04.001.
- [Background] El Sayed MJ, El-Eid GR, Saliba M, Jabbour R, Hitti EA. Improving Emergency Department Door to Doctor Time and Process Reliability: A Successful Implementation of Lean Methodology. Medicine (Baltimore). 2015 Oct;94(42):e1679. doi: 10.1097/MD.0000000000001679. PMID 26496278
- [Background] Patey C, Norman P, Araee M, Asghari S, Heeley T, Boyd S, Hurley O, Aubrey-Bassler K. SurgeCon: Priming a Community Emergency Department for Patient Flow Management. West J Emerg Med. 2019 Jul;20(4):654-665. doi: 10.5811/westjem.2019.5.42027. Epub 2019 Jul 5. PMID 31316707
- [Background] Patey C, Asghari S, Norman P, Hurley O. Redesign of a rural emergency department to prepare for the COVID-19 pandemic. CMAJ. 2020 May 11;192(19):E518-E520. doi: 10.1503/cmaj.200509. Epub 2020 Apr 21. No abstract available. PMID 32317277
- [Background] Killip S, Mahfoud Z, Pearce K. What is an intracluster correlation coefficient? Crucial concepts for primary care researchers. Ann Fam Med. 2004 May-Jun;2(3):204-8. doi: 10.1370/afm.141. PMID 15209195
- [Background] Heaton HA, Castaneda-Guarderas A, Trotter ER, Erwin PJ, Bellolio MF. Effect of scribes on patient throughput, revenue, and patient and provider satisfaction: a systematic review and meta-analysis. Am J Emerg Med. 2016 Oct;34(10):2018-2028. doi: 10.1016/j.ajem.2016.07.056. Epub 2016 Jul 28. PMID 27534432
- [Background] Bellamkonda VR, Kumar R, Scanlan-Hanson LN, Hess JJ, Hellmich TR, Bellamkonda E, Campbell RL, Hess EP, Nestler DM. Pilot Study of Kano "Attractive Quality" Techniques to Identify Change in Emergency Department Patient Experience. Ann Emerg Med. 2016 Nov;68(5):553-561. doi: 10.1016/j.annemergmed.2016.02.005. Epub 2016 Apr 26. PMID 27125817
- [Background] Griffen D, Callahan CD, Markwell S, de la Cruz J, Milbrandt JC, Harvey T. Application of statistical process control to physician-specific emergency department patient satisfaction scores: a novel use of the funnel plot. Acad Emerg Med. 2012 Mar;19(3):348-55. doi: 10.1111/j.1553-2712.2012.01304.x. PMID 22435869
- [Background] Boudreaux ED, Mandry CV, Wood K. Patient satisfaction data as a quality indicator: a tale of two emergency departments. Acad Emerg Med. 2003 Mar;10(3):261-8. doi: 10.1111/j.1553-2712.2003.tb02000.x. PMID 12615592
- [Derived] Rahimipour Anaraki N, Mukhopadhyay M, Patey C, Norman P, Jewer J, Etchegary H, Hurley O, Walsh A, Senior DM, Wang PP, Asghari S. Factors Iinfluencing SurgeCon Implementation in Four Canadian Emergency Departments Guided by Consolidated Framework for Implementation Research. PLoS One. 2025 Dec 2;20(12):e0337389. doi: 10.1371/journal.pone.0337389. eCollection 2025. PMID 41329785
- [Derived] Anaraki NR, Mukhopadhyay M, Jewer J, Patey C, Norman P, Hurley O, Etchegary H, Asghari S. A qualitative study of the barriers and facilitators impacting the implementation of a quality improvement program for emergency departments: SurgeCon. BMC Health Serv Res. 2024 Jul 27;24(1):855. doi: 10.1186/s12913-024-11345-w. PMID 39068432
- [Derived] Mariathas HH, Hurley O, Anaraki NR, Young C, Patey C, Norman P, Aubrey-Bassler K, Wang PP, Gadag V, Nguyen HV, Etchegary H, McCrate F, Knight JC, Asghari S. A Quality Improvement Emergency Department Surge Management Platform (SurgeCon): Protocol for a Stepped Wedge Cluster Randomized Trial. JMIR Res Protoc. 2022 Mar 24;11(3):e30454. doi: 10.2196/30454. PMID 35323121
- [Derived] Anaraki NR, Jewer J, Hurley O, Mariathas HH, Young C, Norman P, Patey C, Wilson B, Etchegary H, Senior D, Asghari S. Implementation of an ED surge management platform: a study protocol. Implement Sci Commun. 2022 Mar 2;3(1):21. doi: 10.1186/s43058-021-00247-1. PMID 35236510
- See also: Canadian Institute for Health Information. Emergency department wait times in Canada continuing to rise — https://www.ipolitics.ca/news/emergency-department-wait-times-on-the-rise-in-canada-cihi-data
- See also: BBC News. Dramatic rise in waiting times at emergency departments — http://www.bbc.com/news/uk-northern-ireland-44562129
- See also: How long is too long to wait in an emergency room? — http://www.huffingtonpost.ca/alan-katz/emergency-room-waits-canada_b_16132058.html
- See also: The Commonwealth Fund. The commonwealth fund 2010 international health policy survey in eleven countries. — http://www.commonwealthfund.org/~/media/files/publications/chartbook/2010/pdf_2010_ihp_survey_chartpack_full_12022010.pdf
- See also: CBC News. Labrador senior waits 10 hours in emergency room without care for broken arm. — http://www.cbc.ca/news/canada/newfoundland-labrador/goose-bay-emergency-wait-time-1.4582333
- See also: CBC News. Picture of senior waiting for hours in St. John's emergency room sparks outrage. — http://www.cbc.ca/news/canada/newfoundland-labrador/senior-hsc-waiting-social-media-1.4587954
- See also: CBC News. St. Anthony patients kept on stretchers while beds remained in storage. — http://www.cbc.ca/news/canada/newfoundland-labrador/hospital-bed-closure-st-anthony-1.4673014
- See also: Canadian Institute for Health Information. PROMS background document. — http://www.cihi.ca/en/patient-experience
- See also: Canadian Institute for Health Information. Patient experience — http://www.cihi.ca/en/patient-experience
- See also: Lean Production. Kaizen — http://www.leanproduction.com/kaizen.html